CLINICAL TRIAL: NCT02698384
Title: Optimisation of Therapeutic Strategies in Acromegalic Subjects Treated With Lanreotide 120mg
Brief Title: Therapeutic Strategies in Acromegalic Subjects Treated With Lanreotide 120mg
Acronym: ACRO-OPTIM
Status: Terminated | Type: Observational
Why Stopped: The study was terminated early due to insufficient potential for recruitment.
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: A-54-52030-315
Record Dates: First submitted 2016-02-26; First posted 2016-03-03 (Estimated); Last update posted 2018-12-21 (Actual); Status verified 2018-12

CONDITIONS: Acromegaly
MeSH Terms: conditions — Acromegaly

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The study aims to evaluate the biochemical and clinical effectiveness on symptoms and tumor size of a monotherapy with Lanreotide 120mg in acromegalic subjects, to describe criteria for starting alternative strategies, and to describe the modalities and the global effectiveness of alternative strategies.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 years or more, suffering from acromegaly
* Treatment naïve or treated subject (whatever the previous treatments except Lanreotide 120mg and radiotherapy) who does not achieve biochemical control in the physician's opinion. Requiring a treatment with Somatostatin analog (SSA)
* Having performed a Magnetic Resonance Imaging (MRI) to evaluate the tumor size within the previous 12 weeks (post-surgery MRI for operated subjects)
* In whom the physician has already decided to initiate a treatment with Lanreotide 120mg as a monotherapy

Exclusion Criteria:

* Subject previously/currently treated with Lanreotide 120mg
* History of radiotherapy for acromegaly
* Subject who requires a surgical intervention for relief of any sign or symptom associated with tumor compression
* Concomitant prolactin hypersecretion requiring a treatment with dopaminergic agonists
* Active neoplastic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acromegalic subjects
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2016-01; Primary Completion 2016-01 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects who achieve a safe concentration of random Growth Hormone (GH) (≤2.5 ng/mL) and normal age and sex-matched Insulin-like Growth Factor-1 (IGF-1) concentration of the monotherapy phase. | Month 5

SECONDARY OUTCOMES:
Profile of subjects | Baseline
  Description of demographics, Patient-Assessed Acromegaly Symptom Questionnaire (PASQ) clinical score, PASQ overall health status, tumor volume, comorbidities, GH and IGF-1 levels
History of acromegaly | Baseline
  Description of the date of diagnosis, GH and IGF-1 levels and tumor volume at diagnosis
History of treatment | Baseline
  Description between the diagnosis of acromegaly and the 1st injection of Lanreotide 120mg (treatments, doses)
Achievement of safe concentration of random GH (≤2.5 ng/mL) and normal age- and sex-matched IGF-1 concentrations of the monotherapy phase | Month 12 and 18
Raw values at each visit and change from baseline in random Growth Hormone (GH) | Baseline, month 5, 12 and 18
Raw values at each visit and change from baseline in overall health status (Patient-Assessed Acromegaly Symptom Questionnaire - PASQ) of the monotherapy phase | Baseline, month 5, 12 and 18
Raw values at each visit and change from baseline in the Acromegaly Quality of Life Questionnaire (ACROQoL total score and each dimension) of the monotherapy phase | Baseline, month 5, 12 and 18
Description of the GH and Insulin-like Growth Factor-1 (IGF-1) levels when the physician decides to start the first alternative strategy | Day 1 (Visit 5)
  Assessed in the alternate strategy phase
Proportion of subjects achieving biochemical control (random GH ≤2.5 ng/mL and normal age- and sex-matched IGF-1 concentrations) at month 18 time point of the alternative strategy phase (18 months after the start of the first alternative strategy) | Month 18
Number of alternative strategies used during the alternative strategy phase | Month 18
Treatments received at least once during the alternative strategy phase | Month 18
Proportion of subjects with clinically relevant tumor shrinkage (tumor volume decrease of ≥ 20% versus V1 (month 0) of the monotherapy phase) at V6 (month 18 time point) of the alternative strategy phase | Month 18
Change in clinical score (PASQ) between baseline (month 0) of the monotherapy phase and month 18 time point of the alternative strategy phase | Month 18
Change in overall health status (PASQ) between baseline (month 0) of the monotherapy phase and month 18 time point of the alternative phase | Month 18
Change in Acromegaly Quality of Life Questionnaire (ACROQoL total score and dimensions) between baseline (month 0) of the monotherapy phase and Month 18 time point of the alternative strategy phase | Month 18

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (10):
- France (10):
  - Hoptial Nord, Amiens
  - Hopital jean Minjoz, Besançon
  - Hopital Neuro-Cardiologique, Fédération d'Endocrinologie, Bron
  - Hopital Albert Michallon, La Tronche
  - Hopital De La Conception, Marseille
  - Hopital Haut Leveque, Pessac
  - Hopital Robert Debre, Reims
  - Hopital Nord, Saint-Etienne
  - Hopital De Hautepierre, Strasbourg
  - Hopital Larrey, Toulouse